CLINICAL TRIAL: NCT04318457
Title: The Application of Response Surface Model on Sedative Endoscopic Retrograde Cholangiopancreatography and Sedative Bronchoscopy
Brief Title: The Application of Response Surface Model on Sedative Procedures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019-01-007BC
Record Dates: First submitted 2020-03-10; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Brochoscopy: 20 ASA Class II-III, aged 20-80 adult patients who require moderate sedation during bronchoscopy will be enrolled into this study. The moderate sedation will be performed only after patients' inform consents and approval of the institutional ethics committee. Patients with conditions such as neurological disorders, hearing impairment, history of habitual sedative medication and alcoholism will be excluded from this study.
- ERCP: 20 ASA Class II-III, aged 20-80 adult patients who require moderate sedation during ERCP will be enrolled into this study. The moderate sedation will be performed only after patients' inform consents and approval of the institutional ethics committee. Patients with conditions such as neurological disorders, hearing impairment, history of habitual sedative medication and alcoholism will be excluded from this study.

SUMMARY:
The purpose of this study is to find the application of Response Surface Model on Sedative Procedures.

DETAILED DESCRIPTION:
It is very important to understand the influence of drug interactions of patients in clinical anesthesia. However, there were only a few quantitative studies on the pharmacodynamics of different drug combinations and patient responses. In recent years, the investigators have innovatively utilized the response surface models in patients receiving painless gastro-intestinal endoscopies. Appropriate pharmacodynamic models of clinical anesthesia for these procedures provide observation, evaluation, and prediction of the pharmacodynamic effects of a combination of clinical anesthetics to such patients. Patients with endoscopic retrograde cholangiopancreatography (ERCP) and bronchoscopy often have a need for painless service, but current clinical studies of using a pharmacodynamic model were lacking in these patients. The investigators therefore design a two-year prospective, observational project to investigate the optimal drug concentration combinations for the shortest wake-up time, adequate analgesia, and appropriate depth of anesthesia for sedative endoscopic ERCP and sedative bronchoscopy using pharmacodynamic models. Multidimensional surface charting will be performed by inputting diversified parameters to predict the drug interactions of the model groups. In this prospective, observational study, the investigators plan to enroll 40 ASA Class Forty ASA Class II-III, aged 20-80 adult patients who require sedative ERCP and bronchoscopy. Moderate to heavy sedation will be performed only after patients' inform consents and approval of the institutional ethics committee. The investigators plan to complete this series of studies within two years: The first year: ERCP(10 patients) and broncoscopy (10 patients). The second year: ERCP(10 patients) and broncoscopy (10 patients). Using response surface models, this study will offer us novel information about patients during procedures which may substantially increase the anesthesia quality and outcome of sedative ERCP and broncoscopy. Physiological signals such as anesthesia depth, drug concentrations and dosages, alertness/sedation score, heart rate, blood pressure, peripheral oxygen saturation, and physical activity responses during painless procedures will be collected and then the above data will be applied to the response surface models. Then the investigators will find the most appropriate anesthetic response surface which may delineate the effects of drug combinations, and will further improve the anesthesia safety and quality for painless ERCP and bronchoscopy patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA Class II-III,
* Aged 20-80 adult patients
* Undergoing moderate sedation during ERCP (endoscopic retrograde cholangiopancreatography) and brochoscopy

Exclusion Criteria:

* Neurological disorders
* Hearing impairment
* History of habitual sedative medication
* Alcoholism

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA Class II-III, aged 20-80 adult patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-03-23 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Response Surface Models | 10 seconds from once the anesthetics were terminated to 10 minutes after the time of each patient's wake up
  Pharmacodynamic response surface model is a mathematic model which provides information about when and what extent the patient will response to a specific physiological condition (pain, respiratory depression, anesthesia depth….) in a given combination drug concentration pairs. The calculated plasma or effect concentration of specific medications will be used to train iteratively by non-linear regression to find the optimal parameters to construct a new response surface model. Then the model will be validated by the observation data to see the accuracy and efficacy of the model.
Evaluation of Response Surface Model Predictions | 10 seconds from once the anesthetics were terminated to 10 minutes after the time of each patient's wake up
  Model predictions were evaluated at the emergence period of moderate sedation or general anesthesia. Model predictions of OAA/S ranging from 0% to 100% were made every 10 seconds from once the anesthetics were terminated to 10 minutes after the time of each patient's wake up. Model predictions were compared with observations with graphical and temporal analyses